CLINICAL TRIAL: NCT06614816
Title: Phase III Clinical Trial of Lyophilized Live Attenuated Varicella Vaccine for Children Aged 1-12 Years
Brief Title: Immunogenicity and Safety of a Live Attenuated Varicella Vaccine in Children Aged 1-12 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Jiangsu CDC (Unknown)
Responsible Party: Principal Investigator, Shiyuan Wang, MD, Department of epidemiology and biostatistics, School of public health,, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT057
Record Dates: First submitted 2024-09-08; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Chickenpox Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Live Attenuated Varicella vaccine candidates (Experimental): The test group received the freeze-dried live attenuated VarV developed by Beijing Minhai Biotechnology Co., LTD., which are derived from the Oka strain, cultured and harvested from inoculated MRC-5 human diploid cells inoculated human diploid cells (MRC-5), and then lyophilized with appropriate stabilizers.
  Interventions: Biological: Oka strain varicella attenuated live vaccine
- Marketed Live Attenuated Varicella vaccine (Active Comparator): the active control group received VarV produced by Changchun BCHT Biotechnology Co.,which are derived from the Oka strain, cultured and harvested from inoculated MRC-5 human diploid cellsinoculated human diploid cells (MRC-5), and then lyophilized with appropriate stabilizers.
  Interventions: Biological: Oka strain varicella attenuated live vaccine

INTERVENTIONS:
Biological: Oka strain varicella attenuated live vaccine — lyophilized powder, subcutaneous injection

SUMMARY:
Immunogenicity and Safety of a Live Attenuated Varicella Vaccine in Children Aged 1-12 Years: A Phase III, Randomized, Double-Blind, Active-Controlled Study

ELIGIBILITY:
Inclusion Criteria:

* Ages ranging from 1 to 12 years for the general healthy population ;
* Obtain informed consent from the volunteer and/or their legal guardian, and sign the informed consent form;
* The volunteer and/or their legal guardian is able to comply with the requirements of the clinical trial protocol;
* Axillary body temperature ≤37.0℃.

Exclusion Criteria:

* Those who have previously been vaccinated against varicella, have a history of varicella or herpes zoster infection;
* Allergy to known components of the study vaccine, or a history of severe allergic reactions to any vaccination;
* A history of epilepsy, seizures, or convulsions, or a family history of psychiatric disorders;
* Individuals with immunodeficiency, undergoing immunosuppressive therapy (e.g., oral corticosteroids), or HIV-related immunocompromised individuals, or those with family members closely exposed to congenital immune diseases;
* Those with congenital malformations, developmental disorders, or severe chronic diseases (such as Down syndrome, diabetes, sickle cell anemia, neurological disorders, Guillain-Barré syndrome);
* Known or suspected concurrent diseases, including respiratory diseases, acute infections, or active chronic diseases, cardiovascular diseases, skin diseases, severe hypertension, or during treatment for malignant tumors;
* Diagnosed with coagulation dysfunction (e.g., deficiency of coagulation factors, coagulation disorders, platelet abnormalities) or significant bruising or coagulation disorders;
* Receipt of blood products within the past 3 months;
* Receipt of attenuated live vaccines within the past 14 days or subunit or inactivated vaccines within the past 7 days;
* Acute illnesses or acute exacerbations of chronic diseases in the past 7 days;
* A history of high fever (axillary body temperature ≥38.0℃) within the past 3 days;
* Any other factors deemed by the investigator as unsuitable for participation in the clinical trial.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
seroconversion rate | 42 days after completing the full course of vaccination.
  The primary immunogenicity endpoint was the seroconversion rate of VZV antibodies

SECONDARY OUTCOMES:
geometric mean titer (GMT) | 42 days after completing the full course of vaccination.
  geometric mean titer (GMT) of VZV antibodies 42 days after vaccination
geometric mean fold increase (GMFI) | 42 days after completing the full course of vaccination.
  geometric mean fold increase (GMFI) of VZV antibodies 42 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Huaiyin District Center for Disease Control and Prevention, Huaian, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No